CLINICAL TRIAL: NCT05896345
Title: Shockwave Lithotripsy (SWL) Versus SWL and Oral Dissolution Therapy (ODT) For Paediatrics Radiolucent Renal Stone. A Randomised Controlled Trial
Brief Title: Shockwave Lithotripsy (SWL) Versus SWL and Oral Dissolution Therapy (ODT) For Paediatrics Radiolucent Renal Stone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Paediatrics RLS
Record Dates: First submitted 2023-05-31; First posted 2023-06-09 (Actual); Last update posted 2023-06-09 (Actual); Status verified 2023-05

CONDITIONS: Pediatric Kidney Disease

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- SWL (Active Comparator): Shockwave Lithotripsy (SWL)
  Interventions: Device: SWL
- SWL and ODT (Active Comparator): Shockwave Lithotripsy (SWL) and Oral Dissolution Therapy (ODT)
  Interventions: Combination Product: SWL and ODT

INTERVENTIONS:
Device: SWL — Shockwave Lithotripsy (SWL) For Paediatrics Radiolucent Renal Stone
  Arms: SWL
Combination Product: SWL and ODT — Shockwave Lithotripsy (SWL) and Oral Dissolution Therapy (ODT) For Paediatrics Radiolucent Renal Stone
  Arms: SWL and ODT

SUMMARY:
To conduct a RCT comparing SWL versus combined ODT and SWL as non-invasive methods for management of paediatrics radiolucent renal stone.

ELIGIBILITY:
Inclusion Criteria:

* 1-2.5 cm renal stone
* Normal Serum creatinine
* Radiolucent stone with Hounsfield units less than 400

Exclusion Criteria:

* Bleeding diatheses.
* Patients with a pacemaker.
* uncontrolled UTIs.
* Severe skeletal malformations.
* Arterial aneurysm in the vicinity of the stone.
* Anatomical obstruction distal to the stone.

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 76 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2021-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Assess the stone free rate measured by computed tomograghy as asymptomatic insignificant residual fragments less than 3 mm | 3 month
  percentage of patient who are stone free

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology Center, Al Mansurah, Outside U.S./Canada, Egypt

IPD SHARING:
Plan to Share IPD: No